CLINICAL TRIAL: NCT06929481
Title: Screening With Liquid Biopsies to Address Colorectal Cancer Inequities
Brief Title: Screening With a DNA Blood Test to Address Colorectal Cancer Inequities
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: CUREBOUND, INC. (Unknown); Family Health Centers of San Diego (Other)
Responsible Party: Principal Investigator, Samir Gupta, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 811489; 316051-00001 (Other Grant/Funding Number: CUREBOUND, INC.)
Record Dates: First submitted 2025-03-16; First posted 2025-04-16 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer Screening; Colorectal Cancer (CRC)
Keywords: cfDNA; cell free DNA blood test; CRC screening; colorectal cancer screening; colorectal cancer inequities; Family Health Centers of San Diego; FHCSD; Guardant Health
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Hematologic Tests; Colonoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Group (Experimental): Participants randomized to the intervention group will be offered expanded colorectal cancer screening options: at home FIT, colonoscopy, or additional option of an in clinic FDA-approved cfDNA blood test with at home FIT.
  Interventions: Device: Cell free DNA (cfDNA) blood test; Other: At home Fecal Immunochemical Test (FIT) or Colonoscopy
- Usual Care Group (Active Comparator): Participants randomized to the usual care group will be offered standard colorectal cancer screening options: at home FIT or colonoscopy.
  Interventions: Other: At home Fecal Immunochemical Test (FIT) or Colonoscopy

INTERVENTIONS:
Device: Cell free DNA (cfDNA) blood test — The intervention is a novel blood test that evaluates circulating cell free tumor DNA (cfDNA) and detects colorectal cancer (CRC). Recently, the cfDNA test has been shown to have 83% sensitivity and 90% specificity for CRC detection, and 13% sensitivity for advanced polyp detection, heralding a new screening strategy postulated to be highly convenient and acceptable. The cfDNA test is made by Guardant Health, FDA approved for average risk colorectal cancer screening, and marketed with the brand name "Shield". Patients opting for the cfDNA test will also be requested to complete an at home FIT.
  Other Names: cfDNA; cfDNA blood test; Guardant Shield cfDNA test; Guardant Shield test
  Arms: Intervention Group
Other: At home Fecal Immunochemical Test (FIT) or Colonoscopy — The usual care group will be offered standard colorectal cancer screening options to choose from: at home FIT or colonoscopy.
  Other Names: at home FIT or colonoscopy

SUMMARY:
Colorectal cancer (CRC) screening participation is suboptimal and associated with inequities in CRC outcomes by race/ethnicity and socioeconomic position. A novel, cell free DNA (cfDNA) blood test has potential to increase participation, but has not been studied in groups at highest risk for adverse CRC outcomes. Among patients age-eligible for colorectal cancer screening, not up-to-date, we propose a 2-arm, pragmatic, randomized controlled trial comparing offers of standard screening options (at home fecal immunochemical test (FIT) or colonoscopy) vs. offers of expanded options (at home FIT, colonoscopy, or in clinic cfDNA plus at home FIT), set at a large Federally Qualified Health Center serving individuals at increased risk for inequities in CRC outcomes. Results will inform guideline and policy makers on whether cfDNA should be supported as a screening option, and support planning for a large-scale trial examining impact of a cfDNA option for screening on CRC and advanced neoplasia detection.

DETAILED DESCRIPTION:
Patients assigned to usual care will be offered options for screening using a standardized script outlining: 1) importance of screening; 2) option of screening with at home FIT or colonoscopy, including key characteristics. Description of key characteristics will include 1) test completion steps; 2) test performance, stating that colonoscopy picks up 9 out of 10 colorectal cancers and important growths called polyps, and that FIT picks up 3 in 4 cancers and 1 in 4 important polyps (we define "important polyps" as adenomas 1 centimeter or larger in size or containing villous/tubulovillous histology or high-grade dysplasia). The script will note abnormal FIT requires a colonoscopy to check for CRC and important growths. Patients assigned to the intervention group will receive an identical offer, but with additional option of screening with an in clinic cfDNA plus an at home FIT. The script will state cfDNA is a blood test meant to be complementary to current screening with ability to detect 8 out of 10 CRCs and 1 in 10 important polyps, and offers advantage of having a same day test for CRC detection to complement the FIT that they will do at home. The script will also state colonoscopy is required if either cfDNA or FIT is abnormal. For patients who opt for the cfDNA plus at home FIT option, the study team will coordinate same day blood draw. Following manufacturer's instructions, 40 mL of blood (4 tubes each with 10 mL of blood) will be collected and sent to Guardant Health for the Guardant Shield test. Patients will be instructed to complete the FIT as soon as possible and within 5 days, and, to minimize the influence of cfDNA result on likelihood of FIT completion, cfDNA results will not be disclosed to the patient for 14 days after the clinic visit. For all subjects, demographic characteristics, coded data on primary provider of record, and outcomes will be collected. Because this is planned as a pragmatic trial to mimic the potential impact of introducing the cfDNA test into usual care, and because the study poses minimum risk and promotes potentially lifesaving colorectal cancer screening, a waiver of informed consent for study screening and randomization to study group assignment, and for written documentation of informed consent has been approved. An informed consent sheet with the option to "opt out" of the study will be provided to all potential subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Persons, aged 45 to 75 years old
2. Not up-to-date with screening, defined based on an existing electronic health record (EHR)-based flag that indicates absence of FIT within the last 12 months, colonoscopy within the last 10 years, sigmoidoscopy within the last 5 years or multi-target stool DNA (Cologuard) test within 3 years.
3. Attending primary care visits during the 2 months of recruitment. According to routine practice, screening status will be confirmed by primary care providers as part of routine visits.
4. Being provided the informed consent form.

Exclusion Criteria:

1. Personal history of colorectal cancer (CRC), adenomas, or other related cancers.
2. Prior history of colorectal surgery
3. Family history of CRC, defined as having one or more first-degree relative (parent, sibling, or child) diagnosed with CRC at any age.
4. Up-to-date with colorectal cancer screening, defined as:

   * Fecal occult blood test (FOBT) or FIT within the last 12 months
   * FIT-DNA (Cologuard) or FIT-RNA (Colosense) test within 3 years
   * cfDNA (Shield) within the last year
   * CT colonography within the last 5 years
   * Sigmoidoscopy within the last 5 years
   * Colonoscopy within the last 10 years
5. Abnormal FIT, FOBT, cfDNA, FIT-DNA, or FIT-RNA test within the last 3 years.
6. Personal history of any of the following high-risk conditions for colorectal cancer:

   * Inflammatory Bowel Disease (IBD), including chronic ulcerative colitis (CUC) and Crohn's disease
   * Familial adenomatous polyposis (FAP)
   * Other hereditary cancer syndromes including but not limited to:

     * Hereditary non-polyposis colorectal cancer syndrome (HNPCC) or "Lynch Syndrome", Peutz-Jeghers Syndrome, MUTYH Polyposis (MAP), Familial Adenomatous Polyposis (FAP), Cowden's Syndrome, Juvenile Polyposis, Serrated Polyposis Syndrome
7. Uninsured patients will be excluded because of inability to ensure follow up. Because of recently expanded Medi-Cal eligibility, exclusions due to insurance are expected to be minimal.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Screening completion | 60 Days
  A single primary outcome measure, screening completion within 60 days of enrollment, is planned. The outcome measure will be defined as the proportion of people enrolled who complete a colorectal cancer screening test within 60 days of enrollment. The definition of colorectal cancer screening test completion includes exposure to a fecal immunochemical test, colonoscopy, or cell free DNA test. The outcome measure will be computed for the standard versus expanded option groups, and compared via a chi-squared test of proportions.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Gupta, MD, MSCS, AGAF, Principal Investigator — University of California, San Diego; Job G Godino, PhD, Principal Investigator — Family Health Centers of San Diego
Locations (1):
- Family Health Centers of San Diego, Logan Heights site, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
All IPD collected throughout the trial will only be used for the purposes of statistical analysis, scientific reporting, and publication.

REFERENCES:
- [Background] Gupta S, Halm EA, Rockey DC, Hammons M, Koch M, Carter E, Valdez L, Tong L, Ahn C, Kashner M, Argenbright K, Tiro J, Geng Z, Pruitt S, Skinner CS. Comparative effectiveness of fecal immunochemical test outreach, colonoscopy outreach, and usual care for boosting colorectal cancer screening among the underserved: a randomized clinical trial. JAMA Intern Med. 2013 Oct 14;173(18):1725-32. doi: 10.1001/jamainternmed.2013.9294. PMID 23921906
- [Background] Singal AG, Gupta S, Tiro JA, Skinner CS, McCallister K, Sanders JM, Bishop WP, Agrawal D, Mayorga CA, Ahn C, Loewen AC, Santini NO, Halm EA. Outreach invitations for FIT and colonoscopy improve colorectal cancer screening rates: A randomized controlled trial in a safety-net health system. Cancer. 2016 Feb 1;122(3):456-63. doi: 10.1002/cncr.29770. Epub 2015 Nov 4. PMID 26535565
- [Background] Gupta S, Miller S, Koch M, Berry E, Anderson P, Pruitt SL, Borton E, Hughes AE, Carter E, Hernandez S, Pozos H, Halm EA, Gneezy A, Lieberman AJ, Sugg Skinner C, Argenbright K, Balasubramanian B. Financial Incentives for Promoting Colorectal Cancer Screening: A Randomized, Comparative Effectiveness Trial. Am J Gastroenterol. 2016 Nov;111(11):1630-1636. doi: 10.1038/ajg.2016.286. Epub 2016 Aug 2. PMID 27481306
- [Background] Singal AG, Gupta S, Skinner CS, Ahn C, Santini NO, Agrawal D, Mayorga CA, Murphy C, Tiro JA, McCallister K, Sanders JM, Bishop WP, Loewen AC, Halm EA. Effect of Colonoscopy Outreach vs Fecal Immunochemical Test Outreach on Colorectal Cancer Screening Completion: A Randomized Clinical Trial. JAMA. 2017 Sep 5;318(9):806-815. doi: 10.1001/jama.2017.11389. PMID 28873161
- [Background] Lieberman A, Gneezy A, Berry E, Miller S, Koch M, Ahn C, Balasubramanian BA, Argenbright KE, Gupta S. Financial Incentives to Promote Colorectal Cancer Screening: A Longitudinal Randomized Control Trial. Cancer Epidemiol Biomarkers Prev. 2019 Nov;28(11):1902-1908. doi: 10.1158/1055-9965.EPI-19-0039. Epub 2019 Aug 6. PMID 31387970
- [Background] Lieberman A, Gneezy A, Berry E, Miller S, Koch M, Argenbright KE, Gupta S. The effect of deadlines on cancer screening completion: a randomized controlled trial. Sci Rep. 2021 Jul 6;11(1):13876. doi: 10.1038/s41598-021-93334-1. PMID 34230556
- [Background] Castaneda SF, Gupta S, Nodora JN, Largaespada V, Roesch SC, Rabin BA, Covin J, Ortwine K, Preciado-Hidalgo Y, Howard N, Halpern MT, Martinez ME. Hub-and-Spoke centralized intervention to optimize colorectal cancer screening and follow-up: A pragmatic, cluster-randomized controlled trial protocol. Contemp Clin Trials. 2023 Nov;134:107353. doi: 10.1016/j.cct.2023.107353. Epub 2023 Oct 5. PMID 37802222
- [Background] Arredondo EM, Dumbauld J, Milla M, Madanat H, Coronado GD, Haughton J, Garcia-Bigley F, Ramers C, Nodora J, Bharti B, Lopez G, Diaz M, Marquez J, Gupta S. A Promotor-Led Pilot Study to Increase Colorectal Cancer Screening in Latinos: The Juntos Contra El Cancer Program. Health Promot Pract. 2021 Jul;22(4):491-501. doi: 10.1177/1524839920912240. Epub 2020 Mar 22. PMID 32202155
- [Background] De La Torre CL, Dumbauld JN, Haughton J, Gupta S, Nodora J, Giacinto RE, Ramers C, Bharti B, Wells K, Lopez J, Diaz M, Moody J, Arredondo EM. Development of a Group-Based Community Health Worker Intervention to Increase Colorectal Cancer Screening Among Latinos. Hisp Health Care Int. 2021 Mar;19(1):47-54. doi: 10.1177/1540415320923564. Epub 2020 May 29. PMID 32466687
- [Background] Castaneda SF, Bharti B, Rojas M, Mercado S, Bearse AM, Camacho J, Lopez MS, Munoz F, O'Connell S, Liu L, Talavera GA, Gupta S. Outreach and Inreach Strategies for Colorectal Cancer Screening Among Latinos at a Federally Qualified Health Center: A Randomized Controlled Trial, 2015-2018. Am J Public Health. 2020 Apr;110(4):587-594. doi: 10.2105/AJPH.2019.305524. Epub 2020 Feb 20. PMID 32078353
- [Background] Bharti B, May FFP, Nodora J, Martinez ME, Moyano K, Davis SL, Ramers CB, Garcia-Bigley F, O'Connell S, Ronan K, Barajas M, Gordon S, Diaz G, Ceja E, Powers M, Arredondo EM, Gupta S. Diagnostic colonoscopy completion after abnormal fecal immunochemical testing and quality of tests used at 8 Federally Qualified Health Centers in Southern California: Opportunities for improving screening outcomes. Cancer. 2019 Dec 1;125(23):4203-4209. doi: 10.1002/cncr.32440. Epub 2019 Sep 3. PMID 31479529
- [Background] Mohl JT, Ciemins EL, Miller-Wilson LA, Gillen A, Luo R, Colangelo F. Rates of Follow-up Colonoscopy After a Positive Stool-Based Screening Test Result for Colorectal Cancer Among Health Care Organizations in the US, 2017-2020. JAMA Netw Open. 2023 Jan 3;6(1):e2251384. doi: 10.1001/jamanetworkopen.2022.51384. PMID 36652246
- [Background] Ciemins EL, Mohl JT, Moreno CA, Colangelo F, Smith RA, Barton M. Development of a Follow-Up Measure to Ensure Complete Screening for Colorectal Cancer. JAMA Netw Open. 2024 Mar 4;7(3):e242693. doi: 10.1001/jamanetworkopen.2024.2693. PMID 38526494
- [Background] Shareef F, Bharti B, Garcia-Bigley F, Hernandez M, Nodora J, Liu J, Ramers C, Nery JD, Marquez J, Moyano K, Rojas S, Arredondo E, Gupta S. Abnormal Colorectal Cancer Test Follow-Up: A Quality Improvement Initiative at a Federally Qualified Health Center. J Prim Care Community Health. 2024 Jan-Dec;15:21501319241242571. doi: 10.1177/21501319241242571. PMID 38554066
- [Background] Ladabaum U, Mannalithara A, Weng Y, Schoen RE, Dominitz JA, Desai M, Lieberman D. Comparative Effectiveness and Cost-Effectiveness of Colorectal Cancer Screening With Blood-Based Biomarkers (Liquid Biopsy) vs Fecal Tests or Colonoscopy. Gastroenterology. 2024 Jul;167(2):378-391. doi: 10.1053/j.gastro.2024.03.011. Epub 2024 Mar 26. PMID 38552670
- [Background] Lieberman DA; AGA CRC Workshop Panel. Commentary: Liquid Biopsy for Average-Risk Colorectal Cancer Screening. Clin Gastroenterol Hepatol. 2024 Jun;22(6):1160-1164.e1. doi: 10.1016/j.cgh.2024.01.034. Epub 2024 Mar 26. No abstract available. PMID 38552672
- [Background] Coronado GD, Jenkins CL, Shuster E, Johnson C, Amy D, Cook J, Sahnow S, Zepp JM, Mummadi R. Blood-based colorectal cancer screening in an integrated health system: a randomised trial of patient adherence. Gut. 2024 Mar 7;73(4):622-628. doi: 10.1136/gutjnl-2023-330980. PMID 38176899
- [Background] Chung DC, Gray DM 2nd, Singh H, Issaka RB, Raymond VM, Eagle C, Hu S, Chudova DI, Talasaz A, Greenson JK, Sinicrope FA, Gupta S, Grady WM. A Cell-free DNA Blood-Based Test for Colorectal Cancer Screening. N Engl J Med. 2024 Mar 14;390(11):973-983. doi: 10.1056/NEJMoa2304714. PMID 38477985
- [Background] Siegel RL, Wagle NS, Cercek A, Smith RA, Jemal A. Colorectal cancer statistics, 2023. CA Cancer J Clin. 2023 May-Jun;73(3):233-254. doi: 10.3322/caac.21772. Epub 2023 Mar 1. PMID 36856579